CLINICAL TRIAL: NCT02237781
Title: Prospective Randomized Trial on the Level of Anti-Mullerian Hormone (AMH) in Women Undergoing Controlled Ovarian Stimulation for IVFwith Gonadotropins.
Brief Title: Levels of Anti-Mullerian Hormone (AMH) During Ovarian Stimulation With Gonadotropins
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Athens (Other)
Collaborators: Lito Maternity Hospital (Other)
Responsible Party: Principal Investigator, Nikos Vlahos, Associate Professor of Obstetrics and Gynecology, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV24042014
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Female Infertility
Keywords: AMH; IVF; ovarian stimulation
MeSH Terms: conditions — Infertility, Female | interventions — Gonadotropins; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMH levels (Experimental): Patients in this group will be stimulated according to a short stimulation protocol with gonadotropins and GnRH antagonists. Levels of AMH will be measured prior and during the ovarian stimulation.
  Interventions: Drug: Gonadotropins

INTERVENTIONS:
Drug: Gonadotropins — The dose of gonadotropins either in the form of a combination of highly purified urinary FSH and LH or with a combination of Rec FSH and Rec LH will depend on the levels of E2 and FSH prior to ovarian stimulation .
  Other Names: Menopure; Gonal

SUMMARY:
Anti-Mullerian Hormone (AMH) is produced only in small ovarian follicles with quite stable levels during the cycle. There is not yet sufficient data to inform couples undergoing IVF about the effect of ovarian stimulation on the levels of AMH due to the increasing size of follicles and chances of success of the method.

DETAILED DESCRIPTION:
Patients undergoing IVF will be included in the study. All patients will be counseled regarding their prognosis. Anti-Mullerian Hormone (AMH) will be measured prior to the initiation of IVF and during ovarian stimulation. Patients will be stimulated with a short GnRH-antagonist protocol. All women will have measurements of serum FSH and estradiol (E2) and a pelvic sonogram on the second day of their cycle. Ovarian stimulation will be initiated with of gonadotropins either in the form of a combination of highly purified urinary FSH and LH or with a combination of Rec FSH and Rec LH. The dose of gonadotropins will depend on the levels of estradiol and FSH prior stimulation. All patients will be re-evaluated on day 3 and 5 of the stimulation (measurment of AMH, E2 and pelvic sonogram), and dosage adjustments will be made and the antagonists (Cetrorelix or ganirelix 0.25 mg/day) will be initiated on day 5. Measurment of AMH, E2 and pelvic sonogram to conferm the size of follicles will be continue every second day untill the oocyte retrieval. When at least 2 follicles reach an average diameter of 17 mm, final oocyte maturation will be triggered with 10,000IU of hCG ( Pregnyl, Organon, Greece Inc.). Oocyte retrieval will be performed 34 to 36 hours later. Patients with successful fertilization will have embryo transfer under sonographic guidance on day 3 after retrieval.

ELIGIBILITY:
Inclusion Criteria:

* All infertile women undergoing ovarian stimulation for IVF.

Exclusion Criteria:

* Women who can not undergo IVF

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Level of AMH | 6 months
  Anti-Mullerian Hormone (AMH) will be measured prior to the initiation of treatment and during ovarian stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Vlahos, MD, Principal Investigator — University of Athens, 2nd Department of Obstetrics and Gynecology